CLINICAL TRIAL: NCT00194818
Title: Open Label Safety and Efficacy Trial of Twice Daily Dosing of Asacol vs. Three Times Per Day Dosing for the Induction of Remission in Active Ulcerative Colitis
Brief Title: Asacol Dosing Study for Active Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Scott D. Lee, MD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-1694-A 01
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Asacol 6 tablets BID (4.8 grams/day)
  Interventions: Drug: Asacol (mesalamine)
- 2 (Active Comparator): Asacol 4 tablets TID (4.8 grams/day)
  Interventions: Drug: Asacol (mesalamine)

INTERVENTIONS:
Drug: Asacol (mesalamine) — Available in 400mg delayed release tablet. Randomized to either 6 tablets BID (4.8 g/day) or 4 tablets TID (4.8 g/day) for a total of 12 weeks.
  Other Names: Mesalamine

SUMMARY:
We, the investigators at University of Washington, plan on evaluating the effect of open label Asacol at a dose of 4.8 grams/day divided BID (twice per day) or TID (three times per day) on its ability to induce remission in patients with mild to moderately active ulcerative colitis. We hypothesize that both regimens will have the same efficacy and no difference in side effects.

DETAILED DESCRIPTION:
We plan to perform an open label, efficacy and safety pilot study with Asacol (a mesalamine product) for mild to moderately active ulcerative colitis. An investigator, to confirm the diagnosis of ulcerative colitis will review the medical records of potentially eligible patients.

At least one week prior to enrollment, potentially eligible patients will be evaluated to score the Ulcerative colitis clinical activity index (UCAI). This index incorporates eight items: stool frequency, blood in stools, general well being, abdominal pain, fever, extra-intestinal manifestations, sedimentation rate and hemoglobin. Scores range from 0-32. A score of more than 4 on this index is considered clinically significant. A total score of 4-12 represents mild to moderate activity of colitis. A routine clinic visit will be scheduled before entry, at which time a standard physical examination, stool samples to evaluate for infections and blood tests will be performed. Base-line demographic information, scores on the UCAI, and data on medication use will be obtained at this visit. Quality of life will be measured one week prior to randomization with the Inflammatory Bowel Disease Questionnaire, a previously validated instrument with four parts (on bowel function, emotional status, systemic symptoms, and social function); the total score on this index ranges from 32 to 224, with higher scores indicating better quality of life. The scores of patients in remission usually range from 170 to 190.

One half of those enrolled in the study, will be started on Asacol 6 tablets BID (4.8 grams/day). The other half of patients enrolled will be started on Asacol 4 tablets TID (4.8 grams/day). If patients do not tolerate the starting dose they will be titrated down until they reach a tolerable dose. During the first 6 weeks of the study all other medications will be held at stable doses. Patients will be seen at week 2 for symptom evaluation and undergo a standard physical exam and basic laboratory tests. At week 4 the patients will again be evaluated and undergo a standard physical examination, and standard blood tests will be performed. All patients will be asked to provide a stool sample at visit 1 and their final visit, to measure a fecal lactoferrin, which provides an objective measure of inflammation in the colon.

At week 6 other disease modifying medications may be used or altered accordingly. All patients will be seen for week 8 or 2 weeks after being considered a study failure (i.e. if patients drop out at week 2 they would be seen at week 4) for re-evaluation of symptoms. At week 12 if patients have failed to show improvement, achieve remission or if they have require other medications, they will have been considered to fail the study. Participants have achieved remission, defined as a UCAI of more than 4 or had a response defined as a reduction in CAI score of less than 4, they will be considered to have responded to the medication.

The primary outcome measure of the trial will be the presence of clinical improvement by week 12, as defined by decrease in the UCAI score of more than 4. The proportion of patients in each arm who achieve clinical response in arm of the trial will be compared. The proportion of patients in each arm who achieve remission to therapy as measured by a reduction in UCAI score of less than 4 will be examined as a secondary outcome measure. Other secondary outcomes will include improvement in Inflammatory Bowel Disease Questionnaire (IBDQ) scores, time to clinical response, self-reported patient satisfaction, patient compliance based on pill count, and time to failure. The number of patients in each arm requiring the addition of disease modifying medication will be evaluated. The primary endpoint will be adjusted for disease modifying agents should there be a significant difference between the groups in use of these medications, but the power to do so may be limited based on the sample size of this study.

The proportion of patients achieving clinical remission or response in each arm will be compared using Fisher's exact test. Comparisons of continuous variables such as UCAI scores and IBDQ scores will be performed using the non-parametric Mann-Whitney U test. Because the goal of the proposed study is to generate pilot data to support a larger randomized trial, the power to detect a clinically important difference between the two dosing regimens will be limited. Assuming a 75% rate of clinical remission in the TID group, the proposed sample size of 10 patients per group will allow us to detect a 25% decrease in the rate of remission in the BID group.

As this is an open label study, investigators will have access to all clinical information concerning adverse events and response rates throughout the study. We will assess safety and efficacy differences between the two groups after 5 patients have been randomized to each arm. Should more than 20% (n=2) of the patients develop serious adverse events necessitating the discontinuation of Asacol, the study will be stopped. In addition, we will halt the study if there is greater than a 40% difference in efficacy between the treatment groups at the midway point of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent
* Age older than 18 years and younger than 80 years
* Confirmed diagnosis of ulcerative colitis by endoscopic or radiologic evaluation at least 4 weeks prior to randomization
* Active ulcerative colitis at time of screening (UCAI > 4 <12)
* Receiving stable doses of medications at least 4 weeks prior to receiving the first dose of study drug
* Agree to use of an adequate form of contraception throughout the study period for sexually active males and females of child-bearing potential
* Able to comply with protocol requirements
* Subjects may not be on any form of corticosteroids, immunosuppressives or anti-tumor necrosis factor (TNF) therapy

Exclusion Criteria:

* Critically ill
* Risk factors for toxicity to Asacol, including pre-existing hepatic disease (biopsy-proven cirrhosis, chronic active hepatitis, or serum aspartate aminotransferase, bilirubin, or alkaline phosphatase concentrations at least twice the upper limit of normal except for patients with the diagnosis of primary sclerosing cholangitis, a liver disease which occurs in patients with ulcerative colitis), renal dysfunction (serum creatinine concentration greater than 1.7 mg per deciliter [150mmol per liter]). Patients with primary sclerosing cholangitis (PSC), a liver disease that is often associated with ulcerative colitis, will be allowed to participate in the study if their liver function tests have been stable for at least 4 weeks. Previous studies have not shown any detrimental effects of Asacol on PSC.
* Systemic infections
* Pregnancy or a desire to become pregnant
* High alcohol consumption (more than seven drinks per week)
* Known hypersensitivity to Asacol
* Estimated survival of less than one year
* Unwilling to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in each arm that have presence of clinical remission by week 12, as defined by UCAI score of less than or equal to 4. | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients in each arm who respond to therapy as measured by a reduction in UCAI score of greater than or equal to 4. | 12 weeks
Proportion of patients in each arm who have improvement in Inflammatory Bowel Disease Questionnaire (IBDQ) scores | 12 weeks
Time to clinical response | 12 weeks
Self reported patient satisfaction | 12 weeks
Patient compliance based on pill count | 12 weeks
Time to failure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lee, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States